CLINICAL TRIAL: NCT03730506
Title: Assessment of the Accuracy of Surgical Guide Designed From Digital Impression, Dental Model Scanning Using CBCT and Desktop Scanner in Computer Guided Implantology: Randomized Clinical Trial
Brief Title: Assessment of the Accuracy of Surgical Guide Designed From Digital Impression, Dental Model Scanning Using CBCT and Desktop Scanner in Computer Guided Implantology:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr taha Adu el wafa, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAD2:7:1
Record Dates: First submitted 2018-10-22; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Computer Guided Implant

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBCT (Experimental)
  Interventions: Device: Intra oral scanner
- IOS (Experimental)
  Interventions: Device: Intra oral scanner
- desktop scanner (Active Comparator)
  Interventions: Device: Intra oral scanner

INTERVENTIONS:
Device: Intra oral scanner — computer guided implant
  Other Names: CBCT; desktop scanner

SUMMARY:
Assessment of the Accuracy of Surgical Guide Designed from Digital Impression, Dental Model Scanning using CBCT and Desktop Scanner in Computer Guided Implantology:

Randomized Clinical Trial.

DETAILED DESCRIPTION:
Research question:

In computer guided Implantology, are surgical stents designed from scan of dental model by CBCT and from digital impression as accurate as surgical stents designed from desktop scanner?

Statement of the problem:

The role digital dentistry is improved in computer guided implantology especially with development of computer guided implant software, desktop scanner and intra oral scanner development and CBCT machines.

Intra-oral scanner, desktop scanner and CBCT scanner can be used in creation of 3D digital model that can be used with computer guided implant in fabrication of the surgical stent.

And the question, is the accuracy of surgical guide will be affected when designed by one of these different modalities?

Rationale for conducting the research:

Digital 3D dentoginival details are very important in computer guided implantology and designing of surgical stent.nowadays there are many methods to obtain this soft tissue replica as CBCT,desktop scanner and intra oral scanner.this study is conducted to asses the effect of different method of soft tissue digitization on the accuracy of surgical template used in computer guided implantology.

ELIGIBILITY:
Inclusion Criteria:

* partially edentulous patient.
* Patients with bucco-lingual bone thickness more than 6 mm allowing flapless implant placement.

Exclusion Criteria:

* Completely edentulous patient or Free end saddle edentulous area.
* Patients needing graft or sinus lifting with implant placement.
* Patients with thin ridges.
* Patients with systemic disease that may affect bone quality.
* Patients with poor oral hygiene and active periodontal diseases.
* Patient with limited mouth opening

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of angular deviation of virtual implants and actual implant position by 3rd party software in degrees | one year
  Evaluation of angular deviation of virtual implants and actual implant position by 3rd party software in degrees to assess the accuracy of surgical guide

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT03730506/Prot_000.pdf